CLINICAL TRIAL: NCT07382219
Title: Real-World Effectiveness of Nirsevimab Against RSV-Related and All-Cause Respiratory Tract Infections in Chinese Infants: A Multicenter Cohort Study
Brief Title: Real-World Effectiveness of Nirsevimab Against RSV-Related and All-Cause Respiratory Tract Infections in Chinese Infants
Status: Completed | Type: Observational
Sponsor: Han Tongyan (Other)
Responsible Party: Sponsor-Investigator, Han Tongyan, Chief Physician, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: M20250653
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: RSV Infections; Lower Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — nirsevimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Nirsevimab group: Infants who received Nirsevimab during the study period.
  Interventions: Biological: Nirsevimab
- Control group: Infants with health records established at the same study centers during the study period who were eligible for Nirsevimab but did not receive the immunization.

INTERVENTIONS:
Biological: Nirsevimab — Nirsevimab will be administered as a single intramuscular dose of 50 mg for infants < 5 kg and 100 mg for infants ≥ 5 kg.
  Other Names: Beyfortus
  Groups: Nirsevimab group

SUMMARY:
A multicenter, retrospective cohort study based on clinical data from seven tertiary hospitals in China will be undertaken. The study aims to evaluate the real-world effectiveness of Nirsevimab in preventing Respiratory Syncytial Virus (RSV) infections and all-cause respiratory infections. Clinical records will be used to compare outcomes between infants who received Nirsevimab and a control group. The study focuses on infants aged 0 to 1 year during the RSV season.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of Nirsevimab in preventing RSV-related and all-cause lower respiratory tract infections (LRTI) among infants in a real-world setting.

The target population includes infants aged 0 to 1 year enrolled across seven Chinese tertiary hospitals during the RSV season (September 2024 through April 2025). The study employs a target trial emulation design to compare infants receiving Nirsevimab with a control group of infants who did not receive Nirsevimab.

Outcomes will be assessed over a follow-up period of up to 180 days. Researchers will utilize hospital electronic medical records to identify the incidence of infections, hospitalizations, and admissions to the intensive care unit (ICU). Statistical methods, such as inverse probability of treatment weighting, will be applied to balance the characteristics of the two groups and ensure a valid comparison.

ELIGIBILITY:
Inclusion Criteria:

Infants aged ≤ 1 year (including preterm infants) entering their first RSV season.

Exclusion Criteria:

1. Prior or active RSV infection.
2. Prior RSV immunization (maternal vaccine or monoclonal antibody).

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged ≤ 1 year entering their first RSV season between September 2024 and April 2025
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of RSV-related LRTI hospitalization. | From enrollment up to 180 days.
  Number of participants admitted to the hospital (inpatient care) with a diagnosis of LRTI and a laboratory-confirmed RSV infection (detected by PCR or antigen testing).

SECONDARY OUTCOMES:
Incidence of all-cause LRTI hospitalization. | From enrollment up to 180 days.
  Number of participants admitted to the hospital with a diagnosis of LRTI caused by any pathogen (including RSV, other viruses, or bacteria) or unspecified agents.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Inner Mongolia Maternity and Child Health Care Hospital, Hohhot, Inner Mongolia
  - Women and Children's Hospital, Qingdao, Shandong
  - Beijing Children's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No